

## Power analysis

Since there was no similar study in the literature, assuming we can achieve a moderate effect level (dz=0.7), a power analysis was performed before the study. Accordingly, when at least 19 participants per group were included, that would result in 80% power with %95 confidence level.

## **Descriptive Statistics**

Statistical analysis of the data was performed using the SPSS 22.00 statistical package program. Descriptive statistics are presented by Mean ± Standard Deviation values. Intergroup homogeneity was analysed by the Kolmogorov-Smirnov test. Two groups (NIA and Pilates) were defined for this study.

As a result of the test, two groups were found to be homogeneous in terms of descriptive variables. However, given the number of people in the group, nonparametric statistical analysis methods were used.

## **Statistics for Comparison of Interventions**

The t-test was used for the initial measurements of the groups. The Wilcoxon test was used to analyse intragroup changes, and the Mann Whitney-U test was used to analyse inter-group differences. The significance level was set at p<0.05.